CLINICAL TRIAL: NCT04385368
Title: A Phase III, Randomized, Multicenter, Double-blind, Placebo-controlled Study to Determine the Efficacy of Adjuvant Durvalumab in Combination With Platinum-based Chemotherapy in Completely Resected Stage II-III NSCLC (MERMAID-1)
Brief Title: Phase III Study to Determine the Efficacy of Durvalumab in Combination With Chemotherapy in Completely Resected Stage II-III Non-small Cell Lung Cancer (NSCLC)
Acronym: MERMAID-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D910LC00001; 2020-000556-35 (EudraCT Number)
Record Dates: First submitted 2020-04-30; First posted 2020-05-12 (Actual); Results first posted 2024-08-30 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: NCSLC; Double-blind; PD-L1; MEDI4736; Durvalumab; DFS; OS; MRD+; MRD-; Completely Resected Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — durvalumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double- Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Durvalumab + SoC chemotherapy (Experimental): Intravenous administration of Experimental and Standard of Care Therapy
  Interventions: Drug: Durvalumab + SoC chemotherapy
- Placebo + SoC chemotherapy (Placebo Comparator): Intravenous administration of Placebo and Standard of Care Therapy
  Interventions: Other: Placebo + SoC chemotherapy

INTERVENTIONS:
Drug: Durvalumab + SoC chemotherapy — Experimental Treatment
  Other Names: MEDI4736
  Arms: Durvalumab + SoC chemotherapy
Other: Placebo + SoC chemotherapy — Placebo Comparator
  Other Names: Placebo
  Arms: Placebo + SoC chemotherapy

SUMMARY:
This is a Phase III, randomized, parallel-arm, placebo controlled, double blind, multicenter study assessing the efficacy and safety of durvalumab versus placebo following SoC chemotherapy in patients with completely resected stage II-III NSCLC who are MRD+ post surgery

DETAILED DESCRIPTION:
Patients who have no evidence of disease recurrence confirmed by CT and/or MRI and are confirmed to meet all eligibility criteria will be randomized 1:1 to durvalumab + Standard of care (SoC) chemotherapy or placebo + Standard of care (SoC) chemotherapy arm.

The primary objective of this study is to assess the efficacy of durvalumab +SoC chemotherapy compared to placebo+ SoC chemotherapy as measured by DFS in all patients.

ELIGIBILITY:
Inclusion criteria:

Patients must be capable of giving signed informed consent, which includes a mandatory genetic informed consent and compliance with the requirements and restrictions listed in the informed consent forms (ICFs) and in this protocol. Provision of signed and dated, written ICFs must occur prior to any mandatory study-specific procedures, sampling, and analyses.

In addition to ICF1 and ICF2, patients will provide signed and dated written optional genetic informed consent prior to collection of a sample for optional genetic analysis at the time of second screening (Table 2). This is different from the genetic samples and testing covered by ICF1, which are mandatory for participation in this study.

Criteria and procedures initiated with the signing of ICF1

1. ICF1 must be signed and dated prior to any study procedures and prior to the planned surgical resection of the primary NSCLC, with the exceptions noted below. This consent will cover the study-specific first screening procedures outlined in Table 1.

   Exception: Patients will be permitted to sign ICF1 up to Week 3 (Day 21) postsurgery. Patients identified after Week 3 post-surgery but prior to Week 5 (Day 35) post-surgery may be allowed to sign ICF1 depending on the outcome of the discussion with the study physician. In these cases, a whole blood sample and resected tumor tissue must be collected and sent to the diagnostic lab as soon as possible after ICF1 is signed for development of the personalized panel. A plasma sample must still be collected at Week 3-5 (Day 21-35) post-surgery, even if creation of the personalized panel for MRD detection is delayed.

   Age
2. Age ≥18 years at the time of screening. Sex
3. Male and/or female. Type of patient and disease characteristics
4. Individuals who have diagnosis of histologically confirmed NSCLC (WHO 2015 classification) with resectable (stage II-III) disease (according to IASLC Staging Manual in Thoracic Oncology v8.0). Select (ie, T3N2 or T4N2) stage IIIB patients will be eligible, provided that they are upstaged to T3N2 or T4N2 based on confirmed pathology. Patients who are staged asT3N2 or T4N2 prior to surgery are not eligible.
5. A contrast-enhanced CT or MRI scan of the chest must have been done for surgical planning prior to surgery. It is recommended that patients undergo combined FDG-PET (18F-Fluoro-deoxyglucose positron emission tomography) and CT scan (contrastenhanced or low-dose CT component) in order to rule out detectable extrathoracic, extracranial metastasis and to assess for potential mediastinal lymph node involvement prior to surgery. In the absence of pre-operative FDG-PET CT imaging, pre-operative contrast-enhanced CT imaging or MRI scan must cover liver and adrenal glands. If only CT is available, or FDG-PET reveals suspicious lymph node mediastinal involvement, it is recommended that invasive pre-operative mediastinal staging is performed according to the algorithm of the European Society of Thoracic Surgeons guidelines (algorithm to follow for primary mediastinal staging if only pre-operative CT is available [De Leyn et al 2007], algorithm to follow for primary mediastinal staging when PET-CT is available [De Leyn et al 2014]). It is preferred that imaging occurs within 6 weeks prior to surgery. Brain MRI (preferred) or brain CT with IV contrast is required for complete staging of the tumor.
6. Complete resection of the primary NSCLC is mandatory. The primary tumor must be deemed resectable by a multidisciplinary evaluation that must include a thoracic surgeon certified or trained according to local standards and who performs lung cancer surgery as a significant part of their practice. Surgical resection of the primary NSCLC can occur by open thoracotomy or by video-assisted thoracic surgery (VATS) and resection can be achieved by segmentectomy, lobectomy, sleeve resection, bilobectomy, or pneumonectomy. Patients undergoing wedge resection are not eligible for this study. Note: Patients undergoing segmentectomy must have tumors less than 2 cm in maximum diameter. Where a resection has been extended by means of a wedge resection of an adjacent lobe to ensure complete resection of a tumor at or crossing a fissure between lobes, this is acceptable if surgical margins are clear of disease. Where the resection of a second tumor nodule (eg, a T4 lesion) is undertaken by means of a wedge resection of a separate lobe, then the patient is not eligible.

   At a minimum, the following parameters should be met for a tumor to be declared completely resected:
   1. The surgeon performing the resection should remove all gross disease by the end of surgery. All surgical margins of resection must be macroscopically negative for tumor.
   2. Pathology and/or operative reports must include the examination of at least 2 different mediastinal lymph node (N2) levels, one of which is the subcarinal node-group (level 7) and the second of which is lobe-specific (defined below).

      Note: In the uncommon clinical situation where the surgeon thoroughly examines a mediastinal lymph node level and does not find any lymph nodes, that mediastinal lymph node level may be counted among the minimum 2 required levels. However, the surgeon must clearly document in the operative report or in a separate written statement that the lymph node level was explored and no lymph nodes were present. Normal appearing lymph nodes, if present, must be biopsied or removed. Exploration of nodes must clearly be documented in medical file if not recorded in operative report.

      Note: Lobe-specific lymph node stations are classified based on the location of the primary tumor as follows (based on IASLC 2009 lymph node map terminology [Rusch et al 2009]): Stations 2R and 4R for right upper lobe or middle lobe tumors, stations 4L, 5, and 6 for left upper lobe tumors, stations 8 and 9 for lower lobe tumors of both sides (Adachi et al 2017, Rami-Porta et al 2005).
   3. No extracapsular nodal extension of the tumor is observed in resected mediastinal N2 lymph nodes.

   Note: Extracapsular nodal extension in resected N1 nodes is permitted. Note: The highest mediastinal node resected can be positive for malignancy. Note: Carcinoma-in-situ can be present at the bronchial margin.
7. All patients who enrol in the study prior to surgery must have a pre-surgical plasma sample collected for MRD evaluation. Patients will not be excluded from randomization based on the results of analysing the pre-surgical plasma samples.

   The following criteria must be met prior to signing ICF2:
8. Confirmation of suitable samples of resected tumor tissue and whole blood for WES of tumor and germline DNA, respectively, and creation of Sponsor-approved personalized panel for MRD detection. Tumor tissue and whole blood samples must be provided to the diagnostic laboratory for development of the personalized panel as soon as possible.

   Germline sequencing of whole blood is mandatory. Note: If a patient's tumor has less than the requisite 50 tumor-specific variants, a panel cannot be built and the patient will no longer be able to participate in the study.
9. Established MRD status (MRD+ or MRD-) based on Sponsor-approved personalized assay of a plasma sample collected at Week 3-5 (Day 21-35) post-surgery.
10. Known tumor PD-L1 status determined at a central reference laboratory testing service using a validated Ventana SP263 PD-L1 immunohistochemistry (IHC) assay prior randomization. Patients with unknown PD-L1 status are not eligible for the study.

    Criteria and procedures initiated with the signing of ICF2
11. Post-operative CT scan of the chest (including liver and adrenal glands) performed within 28 days + 7 days prior to randomization. If clinically indicated, additional scans (such as brain MRI [preferred] or brain CT with IV contrast) should be performed to confirm no evidence of metastasis.
12. ICF2 must be signed and dated after MRD status is determined and prior to initiation of any study-specific procedures, sampling, and analyses outlined in SoAs in Table 2 and Table 3. Randomization must occur within the 12 weeks (+ 7 days) following surgery.
13. WHO/Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
14. Complete postoperative wound healing must have occurred prior to randomization; patients must have recovered from all acute, reversible toxic effects from prior treatments (excluding alopecia) that could potentially adversely impact further administration of durvalumab/placebo or chemotherapy according to the Investigator's judgment.
15. Eligible to tolerate 4 cycles of platinum-based adjuvant chemotherapy
16. Adequate organ and marrow function as described in the protocol. 17 Must have a life expectancy of at least 12 weeks Weight 18 Body weight >30 kg

Exclusion criteria:

Diagnostic assessments

1. Post-operative imaging demonstrating unequivocal evidence of disease recurrence or tissue biopsy-proven disease recurrence. In the event of lymphadenopathy on imaging that would lead to exclusion, histopathological confirmation of lymph node metastasis should be obtained prior to excluding a patient from the study. If pathological confirmation of lymph-node metastasis is not technically feasible and imaging appearance are deemed unequivocal for relapse, the patient will be excluded.
2. EGFR-mutant and/or ALK-translocation-positive, as assessed either from a pre-surgical biopsy sample (preferred) or the resected tumor tissue (if biopsy was not evaluable or available). Any of the following scenarios are acceptable for this study:

   Where EGFR/ALK results are obtained from a pre-surgical tissue biopsy as part of standard local practice, the patient must be confirmed EGFR/ALK wild-type prior to enrolling in the study.

   Results obtained from testing the patient's primary tumor tissue during screening for another AstraZeneca study may be used in this study.

   Results from local testing of a pre-surgical biopsy. All local EGFR/ALK testing performed locally must be performed using a well-validated, local regulatory-approved test. EGFR/ALK may be tested centrally if local testing is unavailable. Patients will still be allowed to continue with first screening procedures while testing is ongoing but will not be able to continue into second screening if their tumor tests positive for EGFR mutations and/or ALK translocations.
3. Mixed small cell and NSCLC histology.
4. Require re-resection or are deemed to have unresectable NSCLC by a multidisciplinary evaluation that must include a thoracic surgeon who performs lung cancer surgery as a significant part of their practice.
5. Patients who are candidates to undergo only wedge resections. Medical conditions
6. History of allogeneic organ or bone marrow transplantation.
7. Non-leukocyte-depleted whole blood transfusion within 120 days of genetic sample collection. Note: This exclusion criterion only relates to whole blood and does not include other blood products (eg, packed red blood cells).
8. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [eg, colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:

   * Patients with vitiligo or alopecia
   * Patients with hypothyroidism (eg, following Hashimoto syndrome) stable on hormone replacement
   * Any chronic skin condition that does not require systemic therapy
   * Patients without active disease in the last 5 years may be included but only after consultation with the Study Physician
   * Patients with celiac disease controlled by diet alone
9. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, uncontrolled cardiac arrhythmia, active ILD, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirements, substantially increase risk of incurring AEs, or compromise the ability of the patient to give written informed consent.
10. History of another primary malignancy, except for

    * Malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of IP and of low potential risk for recurrence
    * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
    * Adequately treated carcinoma-in-situ without evidence of disease
11. History of active primary immunodeficiency
12. Active infection, including tuberculosis (clinical evaluation that includes clinical history, physical examination, and radiographic findings, and tuberculosis testing in line with local practice), hepatitis B (HBV; known positive HBV surface antigen [HBsAg] result), hepatitis C (HCV), or human immunodeficiency virus infection (positive HIV 1/2 antibodies). Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for HCV antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
13. Known allergy or hypersensitivity to any of the IPs or any of the IP excipients.
14. Any medical contraindication to treatment with platinum-based doublet chemotherapy as listed in the local labeling.

    Prior/concomitant therapy
15. Received any prior adjuvant therapy for NSCLC or any prior exposure to durvalumab.
16. Any concurrent chemotherapy, IP, biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (eg, hormone replacement therapy) is acceptable.
17. Radiotherapy treatment for NSCLC in the neoadjuvant setting. Radiotherapy treatment to more than 30% of the bone marrow or with a wide field of radiation within 4 weeks of the first dose of IP.
18. Receipt of live attenuated vaccine within 30 days prior to the first dose of IP. Note: Patients, if enrolled, should not receive live vaccine while receiving IP and up to 30 days after the last dose of IP.
19. Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of IP.
20. Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab/placebo. The following are exceptions to this criterion:

    * Intranasal, inhaled, topical steroids, or local steroid injections (eg, intra-articular injection)
    * Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent
    * Steroids as premedication for hypersensitivity reactions (eg, CT scan premedication) Prior/concurrent clinical study experience
21. Participation in another clinical study with an IP administered since completion of surgery.
22. Previous IP assignment in the present study.
23. Concurrent enrollment in another clinical study, unless it is an observational (noninterventional) clinical study, or during the follow-up period of an interventional study.
24. Prior randomization or treatment in a previous durvalumab clinical study regardless of treatment group assignment.

    Other exclusions
25. Patients who are never-smokers; defined as no more than 100 cigarettes or its equivalent in his/her lifetime.
26. Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of durvalumab/placebo.
27. Judgment by the Investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions, and requirements.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2020-07-17 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Solange Peters, Principal Investigator — Centre Hospitalier Universitaire Vaudois (CHUV); Charles Swanton, Principal Investigator — Francis Crick Institute
Locations (125):
- United States (15):
  - Research Site, Birmingham, Alabama
  - Research Site, Long Beach, California
  - Research Site, Santa Rosa, California
  - Research Site, West Hollywood, California
  - Research Site, Miami, Florida
  - Research Site, Silver Spring, Maryland
  - Research Site, Minneapolis, Minnesota
  - Research Site, Lincoln, Nebraska
  - Research Site, Albuquerque, New Mexico
  - Research Site, New York, New York
  - Research Site, Durham, North Carolina
  - Research Site, Spartanburg, South Carolina
  - Research Site, Sioux Falls, South Dakota
  - Research Site, Houston, Texas
  - Research Site, Seattle, Washington
- Research Site, Rosario, Argentina
- Australia (2):
  - Research Site, Camperdown
  - Research Site, St Leonards
- Belgium (5):
  - Research Site, Aalst
  - Research Site, Brussels
  - Research Site, Hasselt
  - Research Site, Leuven
  - Research Site, Roeselare
- Brazil (6):
  - Research Site, Belo Horizonte
  - Research Site, Blumenau
  - Research Site, Fortaleza
  - Research Site, São José do Rio Preto
  - Research Site, São Paulo
  - Research Site, Vitória
- Bulgaria (2):
  - Research Site, Panagyurishte
  - Research Site, Sofia
- Canada (5):
  - Research Site, Victoria, British Columbia
  - Research Site, Saint John, New Brunswick
  - Research Site, Kingston, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
- Czechia (3):
  - Research Site, Olomouc
  - Research Site, Ostrava
  - Research Site, Prague
- Denmark (2):
  - Research Site, Copenhagen
  - Research Site, Odense C
- France (6):
  - Research Site, Bordeaux
  - Research Site, Marseille
  - Research Site, Saint-Herblain
  - Research Site, Strasbourg
  - Research Site, Toulouse
  - Research Site, Villejuif
- Germany (3):
  - Research Site, Esslingen am Neckar
  - Research Site, Gauting
  - Research Site, Regensburg
- Greece (4):
  - Research Site, Athens
  - Research Site, Heraklion
  - Research Site, Holargos, Athens
  - Research Site, Thessaloniki
- Research Site, Hong Kong, Hong Kong
- Hungary (5):
  - Research Site, Budapest
  - Research Site, Gyöngyös - Mátraháza
  - Research Site, Győr
  - Research Site, Szolnok
  - Research Site, Törökbálint
- India (3):
  - Research Site, Bengaluru
  - Research Site, Delhi
  - Research Site, Mohali
- Israel (4):
  - Research Site, Haifa
  - Research Site, Kfar Saba
  - Research Site, Petah Tikva
  - Research Site, Ramat Gan
- Italy (3):
  - Research Site, Meldola
  - Research Site, Orbassano
  - Research Site, Roma
- Japan (10):
  - Research Site, Akashi-shi
  - Research Site, Bunkyō City
  - Research Site, Hiroshima
  - Research Site, Kashiwa
  - Research Site, Kōtoku
  - Research Site, Nagoya
  - Research Site, Osaka
  - Research Site, Sendai
  - Research Site, Sunto-gun
  - Research Site, Yokohama
- Mexico (2):
  - Research Site, Culiacán
  - Research Site, México
- Netherlands (3):
  - Research Site, Breda
  - Research Site, Maastricht
  - Research Site, Zwolle
- Research Site, Lima, Peru
- Poland (5):
  - Research Site, Bydgoszcz
  - Research Site, Gdansk
  - Research Site, Tomaszów Mazowiecki
  - Research Site, Warsaw
  - Research Site, Wroclaw
- Research Site, Floreşti, Romania
- Russia (6):
  - Research Site, Kazan'
  - Research Site, Krasnodar
  - Research Site, Krasnoyarsk
  - Research Site, Moscow
  - Research Site, Novosibirsk
  - Research Site, Saint Petersburg
- Research Site, Singapore, Singapore
- South Korea (3):
  - Research Site, Cheongju-si
  - Research Site, Seoul
  - Research Site, Suwon
- Spain (6):
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Oviedo
  - Research Site, Pamplona
  - Research Site, Santiago de Compostela (A Coruña)
- Research Site, Stockholm, Sweden
- Switzerland (2):
  - Research Site, Lausanne
  - Research Site, Zurich
- Taiwan (4):
  - Research Site, Chiayi City
  - Research Site, Taichung
  - Research Site, Taipei
  - Research Site, Taoyuan District
- Thailand (4):
  - Research Site, Bangkok
  - Research Site, Chiang Mai
  - Research Site, Khon Kaen
  - Research Site, Phisanulok
- Turkey (Türkiye) (4):
  - Research Site, Adana
  - Research Site, Ankara
  - Research Site, Istanbul
  - Research Site, Malatya
- Vietnam (2):
  - Research Site, Hanoi
  - Research Site, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Redacted CSP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D910LC00001&attachmentIdentifier=827e5769-f8cb-4126-a8b8-dfb578a8506f&fileName=D910LC00001_CSP_Redacted.pdf&versionIdentifier=
- See also: Redacted SAP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D910LC00001&attachmentIdentifier=5da584de-0a3e-4be1-b55c-7551572c029f&fileName=D910LC00001_SAP_Redacted.pdf&versionIdentifier=
- See also: Redacted CSR synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D910LC00001&attachmentIdentifier=9873843d-d382-419e-b7cd-835f110c0dbc&fileName=D910LC00001_CSR_Synopsis_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This Phase III, multicenter, randomized, double-blind, placebo-controlled study was conducted in participants with completely resected stage II to III non-small cell lung cancer (NSCLC) at 63 sites across 25 countries from 17 July 2020 to 31 August 2023.
Pre-assignment Details: A total of 89 participants were randomized in a 1:1 ratio to durvalumab given concurrently with standard of care (SoC) chemotherapy followed by durvalumab monotherapy, or to a matched placebo given concurrently with SoC chemotherapy followed by placebo.
Groups:
- Durvalumab + SoC: Participants received durvalumab 1500 milligrams (mg) via intravenous (IV) infusion in combination with SoC chemotherapy on Day 1 of each 3-week cycle for up to 4 cycles, followed by durvalumab monotherapy continued on Day 1 of each 4-week cycle for up to 10 additional cycles until unacceptable toxicity, withdrawal of consent, or another discontinuation criterion was met. For participants with tumors of squamous histology, permitted SoC chemotherapy was a combination of carboplatin (area under the serum drug concentration-time curve [AUC] 6) and paclitaxel 200 milligram per square meter (mg/m^2) via IV infusion on Day 1 of each 3-week cycle, for 4 cycles.
  For participants with tumors of non-squamous tumor histology, permitted SoC chemotherapy regimens were pemetrexed 500 mg/m^2 in combination with either cisplatin 75 mg/m^2 or carboplatin AUC 5, all via IV infusion on Day 1 of each 3-week cycle, for 4 cycles.
- Placebo + SoC: Participants received matching placebo via IV infusion in combination with SoC chemotherapy on Day 1 of each 3-week cycle for up to 4 cycles, followed by matching placebo continued on Day 1 of each 4-week cycle for up to 10 additional cycles until unacceptable toxicity, withdrawal of consent, or another discontinuation criterion was met.
  For participants with tumors of squamous histology, permitted SoC chemotherapy was a combination of carboplatin (AUC 6) and paclitaxel 200 mg/m^2 via IV infusion on Day 1 of each 3-week cycle, for 4 cycles.
  For participants with tumors of non-squamous tumor histology, permitted SoC chemotherapy regimens were pemetrexed 500 mg/m^2 in combination with either cisplatin 75 mg/m^2 or carboplatin AUC 5, all via IV infusion on Day 1 of each 3-week cycle, for 4 cycles.
Period: Overall Study
Arm/Group | Durvalumab + SoC | Placebo + SoC
Started | 45 | 44
Completed | 33 | 36
Not Completed | 12 | 8
Not completed — Death | 5 | 5
Not completed — Physician Decision | 3 | 0
Not completed — Withdrawal by Subject | 4 | 3

BASELINE CHARACTERISTICS:
Population: The Full analysis set (FAS) included all randomized participants.
Groups:
- Durvalumab + SoC: Participants received durvalumab 1500 mg via IV infusion in combination with SoC chemotherapy on Day 1 of each 3-week cycle for up to 4 cycles, followed by durvalumab monotherapy continued on Day 1 of each 4-week cycle for up to 10 additional cycles until unacceptable toxicity, withdrawal of consent, or another discontinuation criterion was met.
  For participants with tumors of squamous histology, permitted SoC chemotherapy was a combination of carboplatin (AUC 6) and paclitaxel 200 mg/m^2 via IV infusion on Day 1 of each 3-week cycle, for 4 cycles.
  For participants with tumors of non-squamous tumor histology, permitted SoC chemotherapy regimens were pemetrexed 500 mg/m^2 in combination with either cisplatin 75 mg/m^2 or carboplatin AUC 5, all via IV infusion on Day 1 of each 3-week cycle, for 4 cycles.
- Total: Total of all reporting groups
Arm/Group | Durvalumab + SoC | Placebo + SoC | Total
Number analyzed (Participants) | 45 | 44 | 89
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.5 (8.78) | 64.5 (7.37) | 65.0 (8.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 15 | 32
  Male | 28 | 29 | 57
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 9 | 18 | 27
  White | 35 | 22 | 57
  Not reported | 1 | 3 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 1 | 5
  Not Hispanic or Latino | 40 | 43 | 83
  Missing | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Disease-free Survival (DFS) in FAS (Using Investigator Assessments According to Response Evaluation Criteria in Solid Tumors 1.1 [RECIST 1.1])
Description: DFS was defined as the time from the date of randomization until either of the following events, whichever occurred first: disease recurrence using Investigator RECIST 1.1 assessments (i.e., local or regional recurrence, distant recurrence, second primary NSCLC) or death from any cause.
Time Frame: Every 12 weeks (q12w) ± 1 week until appearance of RECIST 1.1-defined disease recurrence or until primary DFS analysis, up to 33.28 months
Population: The FAS included all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Durvalumab + SoC | Placebo + SoC
Number analyzed (Participants) | 45 | 44
months | NA [14.062 to NA] — NA indicates that median and upper limit of confidence interval was not estimable due to insufficient number of participants with events at study closure and due to limited duration of follow-up. | NA [21.914 to NA] — NA indicates that median and upper limit of confidence interval was not estimable due to insufficient number of participants with events at study closure and due to limited duration of follow-up.

2. Secondary Outcome: DFS in Minimal Residual Disease-positive (MRD+) Analysis Set (Using Investigator Assessments According to RECIST 1.1)
Description: as for outcome 1
Time Frame: as for outcome 1
Population: The MRD+ analysis set included all participants in the FAS who were MRD+, as determined by results from the post-surgical plasma sample based on the assay that was used at the time of randomization assay.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Durvalumab + SoC | Placebo + SoC
Number analyzed (Participants) | 12 | 11
months | 16.7 [2.661 to NA] — NA indicates that upper limit of confidence interval was not estimable due to insufficient number of participants with events at study closure and due to limited duration of follow-up. | NA [5.585 to NA] — NA indicates that median and upper limit of confidence interval were not estimable due to insufficient number of participants with events at study closure and due to limited duration of follow-up.

3. Secondary Outcome: OS in FAS
Description: OS was defined as the time from the date of randomization until death due to any cause. Any participant not known to have died at the time of analysis was censored based on the last recorded date on which the participant was known to be alive.
Time Frame: From the date of randomization until death due to any cause, up to 35 months
Population: The FAS included all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Durvalumab + SoC | Placebo + SoC
Number analyzed (Participants) | 45 | 44
months | NA [NA to NA] — NA indicates that median, upper and lower limit of confidence interval were not estimable due to insufficient number of participants with events at study closure and due to limited duration of follow-up. | NA [NA to NA] — NA indicates that median, upper and lower limit of confidence interval were not estimable due to insufficient number of participants with events at study closure and due to limited duration of follow-up.

4. Secondary Outcome: Overall Survival (OS) in MRD+ Analysis Set
Description: as for outcome 3
Time Frame: From the date of randomization until death due to any cause, up to 35 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Durvalumab + SoC | Placebo + SoC
Number analyzed (Participants) | 12 | 11
months | NA [9.331 to NA] — NA indicates that median and upper limit of confidence interval were not estimable due to insufficient number of participants with events at study closure and due to limited duration of follow-up. | NA [13.372 to NA] — NA indicates that median and upper limit of confidence interval were not estimable due to insufficient number of participants with events at study closure and due to limited duration of follow-up.

ADVERSE EVENTS:
Time Frame: Treatment emergent adverse events (TEAEs) were collected from first dose of study treatment up to 90 days after the last dose of study treatment, 19.1 months. All-cause mortality was assessed from the start of randomization up to completion of study, 35 months.
Description: The safety analysis set consisted of all randomized participants who received at least 1 dose of study treatment (durvalumab/placebo and/or SoC chemotherapy).
Arm/Group | Durvalumab + SoC | Placebo + SoC
All-Cause Mortality (participants affected / at risk) | 6/45 | 5/44
Serious Adverse Events (participants affected / at risk) | 14/45 | 10/44
Other Adverse Events (participants affected / at risk) | 43/45 | 44/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Durvalumab + SoC (N=45) | Placebo + SoC (N=44)
Pneumonia (Infections and infestations) | 3 (3) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Parkinson's disease (Nervous system disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 2 (2)
Azotaemia (Renal and urinary disorders) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypopituitarism (Endocrine disorders) | 1 (1) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0)
Peripheral artery occlusion (Vascular disorders) | 1 (1) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 3 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 0 (0) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 2 (2)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Durvalumab + SoC (N=45) | Placebo + SoC (N=44)
Nasopharyngitis (Infections and infestations) | 2 (2) | 3 (3)
Urinary tract infection (Infections and infestations) | 3 (3) | 1 (1)
Neutrophil count decreased (Investigations) | 8 (15) | 5 (9)
Platelet count decreased (Investigations) | 3 (5) | 2 (3)
Weight decreased (Investigations) | 2 (2) | 3 (3)
White blood cell count decreased (Investigations) | 7 (10) | 2 (5)
Decreased appetite (Metabolism and nutrition disorders) | 9 (14) | 7 (11)
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 (3) | 3 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (7) | 8 (13)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (6) | 3 (3)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 5 (12)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (3) | 4 (5)
Anosmia (Nervous system disorders) | 3 (3) | 0 (0)
Dizziness (Nervous system disorders) | 4 (4) | 2 (4)
Dysgeusia (Nervous system disorders) | 4 (4) | 2 (4)
Headache (Nervous system disorders) | 8 (9) | 4 (6)
Neuropathy peripheral (Nervous system disorders) | 7 (7) | 5 (5)
Paraesthesia (Nervous system disorders) | 3 (4) | 3 (4)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 6 (6)
Anaemia (Blood and lymphatic system disorders) | 15 (21) | 12 (13)
Insomnia (Psychiatric disorders) | 6 (7) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (9) | 5 (5)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 4 (4)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (5)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Hyperthyroidism (Endocrine disorders) | 6 (6) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 13 (13) | 9 (10)
Dry skin (Skin and subcutaneous tissue disorders) | 4 (4) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (8) | 6 (8)
Rash (Skin and subcutaneous tissue disorders) | 8 (9) | 5 (5)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3)
Hypothyroidism (Endocrine disorders) | 6 (6) | 1 (1)
Hypertension (Vascular disorders) | 3 (3) | 4 (4)
Lacrimation increased (Eye disorders) | 3 (4) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 5 (8) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 5 (6)
Constipation (Gastrointestinal disorders) | 12 (15) | 17 (24)
Diarrhoea (Gastrointestinal disorders) | 11 (15) | 7 (7)
Dry mouth (Gastrointestinal disorders) | 3 (3) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 7 (7)
Nausea (Gastrointestinal disorders) | 19 (32) | 18 (35)
Neutropenia (Blood and lymphatic system disorders) | 8 (10) | 3 (5)
Stomatitis (Gastrointestinal disorders) | 3 (3) | 3 (3)
Vomiting (Gastrointestinal disorders) | 5 (8) | 3 (7)
Asthenia (General disorders) | 7 (10) | 4 (4)
Fatigue (General disorders) | 15 (18) | 12 (13)
Malaise (General disorders) | 1 (4) | 3 (3)
Oedema peripheral (General disorders) | 3 (3) | 3 (3)
Pyrexia (General disorders) | 6 (7) | 2 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 5 (6) | 1 (1)
COVID-19 (Infections and infestations) | 3 (3) | 3 (3)

LIMITATIONS AND CAVEATS:
The sponsor closed enrollment early due to the changes in the treatment landscape. Interpretation of the efficacy results is inconclusive due to the small sample size, resulting in wide confidence intervals, and limited duration of follow-up. The overall safety findings remained consistent with the known safety profiles of durvalumab and SoC chemotherapy. No new safety concerns were identified in this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2022-08-02): https://cdn.clinicaltrials.gov/large-docs/68/NCT04385368/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-15): https://cdn.clinicaltrials.gov/large-docs/68/NCT04385368/SAP_001.pdf